## **COVER PAGE**

# Official Title of the Study:

The Effect of a Project-Based Course on Nursing Students' Critical Thinking, Lifelong Learning, and Individual Innovativeness Skills: A Randomized Controlled Trial

NCT Number (if available):

None

#### **Document Date:**

24 March 2025

# **Principal Investigators**:

Dr. Merve TUNCER, Istanbul University

Dr. Nurten ÖZEN, Istanbul University

## INFORMED CONSENT FORM

You are invited to participate in a research study conducted by Merve TUNCER and Nurten ÖZEN at Istanbul University, titled "The Effect of a Project-Based Course on Nursing Students' Critical Thinking, Lifelong Learning, and Individual Innovativeness Skills: A Randomized Controlled Trial." Participation in this study will take approximately 10 minutes of your time. A total of 38 participants will be included in the study.

The aim of this study is to examine the effect of a project-based course on nursing students' critical thinking, lifelong learning, and individual innovativeness skills. The data collected will be destroyed after the completion of the project on 30/04/2030.

Participation in this study is entirely voluntary. You are expected to respond honestly, without any pressure or influence, and provide answers that reflect your true opinions. Reading and approving this form means you agree to participate in the study. However, you have the right to withdraw from the study at any time, without any consequences.

The information obtained from this study will be used solely for research purposes, and your personal data will be kept confidential. However, your anonymized data may be used for publication purposes. With your permission, your contact information may be shared in a "shared participant pool" to allow other researchers to contact you in the future.

If you need any additional information now or in the future about the purpose of this study, you may contact the researcher, Merve TUNCER, at **mervecaglar90@hotmail.com** or **+90 537 504 8017**. If you would like the general or individual results of the study to be shared with you once the research is complete, please inform the researcher.

Merve TUNCER

Marines

I have read the information provided above, which is required to be given to participants before the study, and I understand the scope and purpose of the study I am invited to participate in, as well as the responsibilities I voluntarily undertake. Both written and verbal explanations about the study were provided by the researcher(s) named below. I have also been verbally informed about the potential risks and benefits of the study. I have been assured that my personal information will be carefully protected.

Under these conditions, I voluntarily agree to participate in the study without any pressure or coercion.

| Participant's: | | |
|----------------------|------|------|
| Full Name: | <br> | <br> |
| Signature: | | |
| Contact Information: | | |
| E-mail: | | |
| Phone Number: | | |